CLINICAL TRIAL: NCT02758262
Title: Effects of Noninvasive Brain Stimulation on Brain Activity and Appetite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2016-478
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hyperphagia
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noninvasive brain stimulation: active (Active Comparator): In active condition, subject will receive stimulation during all the duration of the experimental session.
  Interventions: Device: Noninvasive brain stimulation
- Noninvasive brain stimulation: sham (Placebo Comparator): In sham condition, subject will receive stimulation only at the beginning and at the end of the experimental session.
  Interventions: Device: Noninvasive brain stimulation

INTERVENTIONS:
Device: Noninvasive brain stimulation

SUMMARY:
The goal of this project is to identify brain mechanisms by which Noninvasive brain stimulation (NIBS) could decrease hyperphagia. The investigators will synchronously deliver NIBS and measure brain activity in a randomized, crossover, sham-controlled, fully blind study. This work will reveal brain mechanisms to reduce hyperphagia and may contribute to new therapeutic avenues to treat this eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Hyperphagic

Exclusion Criteria:

* Psychiatric disorders
* Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Food craving assessed by the Food Cravings Questionnaire - State | 1 hour

SECONDARY OUTCOMES:
Brain activity assessed by electroencephalography | 1 hour
Brain activity assessed by blood-oxygen-level dependent contrast imaging | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Centre interdisciplinaire de recherche en réadaptation et intégration sociale, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided